CLINICAL TRIAL: NCT05791201
Title: A Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of VX-264 in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Safety, Tolerability, and Efficacy Study of VX-264 in Participants With Type 1 Diabetes
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX22-264-101; 2024-515583-32-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-264 (Experimental)
  Interventions: Drug: VX-264

INTERVENTIONS:
Drug: VX-264 — Allogeneic human stem cell-derived islets.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and efficacy of VX-264 in participants with type 1 diabetes (T1D).

ELIGIBILITY:
Key Inclusion Criteria:

Clinical history of T1D with greater than or equal to (>=) 5 years duration Participant is on a stable diabetic treatment Consistent use of continuous glucose monitoring (CGM) for at least 4 weeks before Screening and willingness to use CGM for the duration of the study

Key Exclusion Criteria:

Prior islet cell transplant, organ transplant, or cell therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to 24 months
Part B and Part C: Change in Peak C-peptide during Mixed-Meal Tolerance Test (MMTT) | From Baseline and at Day 90

SECONDARY OUTCOMES:
Part C: Change in peak C-peptide during MMTT | From Baseline up to 24 months
Part C: Change in Average Total Daily Insulin Dose | From Baseline up to 24 months
Part C: Proportion of Participants who are Insulin Independent at One Point in Time | From Day 180 up to Day 365
Part C: Change in HbA1c values | From Baseline up to 24 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (6):
  - UHealth Diabetes Research Institute, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Montefiore, Pittsburgh, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
- Canada (4):
  - University of Alberta, Edmonton, Edmonton
  - Montreal Clinical Research Institute, Montreal
  - Toronto General Hospital (TGH), Toronto
  - Vancouver General Hospital, Vancouver
- Dresden Center for Islet Transplantation, Dresden, Germany
- IRCCS Ospedale San Raffaele, Milan, Italy
- Leiden University, Leiden, Netherlands
- Hopiteaux Universitaires de Geneve, Geneva, Switzerland
- United Kingdom (2):
  - Churchill Hospital, Headington
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing